CLINICAL TRIAL: NCT04898218
Title: Effect of Osteoanabolic Exercises on Gait, Balance & Fear of Fall Among Osteoporotic Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Amna Khan, Principal Investigator, Assistant Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amna Khan
Record Dates: First submitted 2020-12-22; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bone Mineral Density; Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Aerobic Exercise Group) (Active Comparator): Warm-up exercises were performed by the participants on a cycle ergometer for a duration of 5-10 minutes. Group A was advised to start walking at a comfortable speed on a treadmill for the duration of 30-60 minutes; the intensity of the exercises was 55-75% of MHR, calculated by using a Karvonen method. Initially with the minimum intensity that was gradually raised up to the intensity of Targeted Heart Rate (THR). Once the THR is achieved the intensity was gradually decelerated and patient proceeded for the cool-down phase for 5-10 min.
  Interventions: Other: Exercise
- Group B (Resistance Exercise Group) (Active Comparator): Group B was instructed for strengthening exercises of ten major muscle groups that include Biceps, Triceps, Pectoralis Major, Deltoid, Latissimus Dorsi, Abdominals, Back Extensors, Hamstrings, Quadriceps and Calf. The intensity of the weight-bearing exercises was calculated using 1 Repetition Maximum (RM) method.
  Interventions: Other: Exercise
- Group C (Osteoanabolic Exercise Group) (Experimental): Group C was performed Osteoanabolic exercise divided into two different phases:
  Aerobic Conditioning Phase Participants were instructed to walk on treadmill for 30-60 min. The intensity of the exercises was 55-75% MHR, calculated by Karvonen method. Intensity gradually raised up to the Targeted Heart Rate (THR). Once the THR is achieved the intensity was gradually decelerated and patient proceeded for the cool-down phase. The participants performed 3 days per week for 12 weeks on alternative days.
  Anaerobic (Resistance) Conditioning Phase Resistance training was started on every alternative day of the aerobic conditioning (3 days per week) for 45 min. The intensity of the weight-bearing exercises was calculated using 1 RM method. Resistance training muscle and protocol was the same as for Group B. The participants performed warm-up and cool down similar to that of group A and group B.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercises were performed for 12 weeks, for the maximum of 6 days/week for Osteoanabolic group, 5 days/week for aerobic group and 3 days/ week for a resistance group as per ACSM, FITT protocol.

SUMMARY:
With the increase in life expectancy women spend more than one-third of their life time in post-menopausal state leading to osteoporosis in later stages. Therefore a decrease in temporal-spatial parameters of gait, high risk of fracture, imbalance in functional parameters, fear of fall and compromised health-related quality of life is observed among osteoporotic females. Several physical activities and balance training programs have been implemented globally but nationally no program has yet been designed catering gait balance and fear of fall altogether as a combined program. Therefore, the aim of this study was to determine the effectiveness of Osteoanabolic exercises on Temporal-Spatial gait parameters, Gait Stability Ratio (GSR) and Bone Mineral Density (BMD) among the osteoporotic females. Moreover, the effectiveness of these exercises was evaluated on dynamic balance using Timed Up and Go Test (TUG).

Furthermore, the impact on fear of fall was identified using Fall Efficacy ScaleInternational (FES-I).

DETAILED DESCRIPTION:
A 3-arm Randomized Controlled Trial was conducted at the Department of Rehabilitation Sciences, Ziauddin Hospital using the envelope method. The participants were screened on the Physical Activity Readiness and You Questionnaire (PARQ &YOU). Ninety-three osteoporotic females were randomly allocated into three groups; where; participant in group A' received aerobic training protocol, a participant in group B' resistance training and participant in group C' Osteoanabolic training. A Frequency Intensity Time Type (FITT) protocol according to the American College of Sports Medicine for aerobic and resistance training was incorporated whereas for Osteoanabolic group combination training protocol was used. Twelve weeks of training was conducted where pre and post readings were calculated using activPAL, TUG, FES-I and Peripheral DXA Scan.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporotic females aged in between 50-75 years
* Not participating in any exercise program for the past 3 months
* Independently ambulatory were included in the study

Exclusion Criteria:

• Red flags that limit the recruitment of participants in an exercise program, for example, vertebral fracture, an unstable heart condition, malignancy

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal osteoporotic females screened through PARQ and YOU
Enrollment: 93 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Gait Velocity | Baseline
  Temporal Spatial Gait Parameter
Gait Velocity | 12 weeks
  Temporal Spatial Gait Parameter
Cadence | Baseline
  Temporal Spatial Gait Parameter
Cadence | 12 weeks
  Temporal Spatial Gait Parameter
Gait Stability Ratio | Baseline
  Temporal Spatial Gait Parameter
Gait Stability Ratio | 12 weeks
  Temporal Spatial Gait Parameter
Balance | Baseline
  Balance was measured through Timed-up and Go Test
Balance | 12 weeks
  Balance was measured through Timed-up and Go Test
Fear of Fall | Baseline
  Measured through Fall Efficacy Scale- International consisting of 16 items that are summed to calculate a total score from minimum 16 to maximum 64. Higher the score, greater the fear of falling.
Fear of Fall | 12 weeks
  Measured through Fall Efficacy Scale- International consisting of 16 items that are summed to calculate a total score from minimum 16 to maximum 64. Higher the score, greater the fear of falling.

SECONDARY OUTCOMES:
Bone Mineral Density | Baseline
  Measured through Peripheral DXA Scan on right side calcaneal bone
Bone Mineral Density | 12 weeks
  Measured through Peripheral DXA Scan on right side calcaneal bone

CONTACTS AND LOCATIONS:
Overall Officials: Amna Khan, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No